CLINICAL TRIAL: NCT05280275
Title: A Phase 1/2, Dose and Schedule Evaluation Study to Investigate the Safety and Clinical Activity of Belantamab Mafodotin Administered in Combination With Daratumumab, Lenalidomide and Dexamethasone in Patients With Newly Diagnosed Multiple Myeloma Transplant Ineligible (EAE 120)
Brief Title: A Study to Investigate the Safety and Clinical Activity of Belantamab Mafodotin in Combination With Daratumumab, Lenalidomide and Dexamethasone in Patients With Newly Diagnosed Multiple Myeloma Transplant Ineligible
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Hellenic Society of Hematology (Other)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: EAE120
Record Dates: First submitted 2022-02-21; First posted 2022-03-15 (Actual); Last update posted 2023-12-01 (Actual); Status verified 2023-11

CONDITIONS: Multiple Myeloma; Neoplasms; Neoplasms, Plasma Cell; Gammopathy, Monoclonal; Paraproteinemias; Blood Protein Disorders; Haematologic Disease; Corneal Disease
MeSH Terms: conditions — Multiple Myeloma; Neoplasms; Neoplasms, Plasma Cell; Paraproteinemias; Blood Protein Disorders; Hematologic Diseases; Corneal Diseases | interventions — daratumumab; Lenalidomide; Dexamethasone

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Part 1: Dose Finding (Experimental): Belantamab mafodotin will be administered as a combination therapy as a calculated dose on Day 1 of every other 28-day cycle.
  Belantamab mafodotin starting dose:
  1. Cohort 1: 1.9 Q8W = 1.9 mg/kg on Day 1 of every other 28-day cycle
  2. Cohort 2: 1.4 Q8W = 1.4 mg/kg on Day 1 of every other 28-day cycle
  Administration schedule for daratumumab 1800mg SC (fixed dose):
  Cycles 1-2: days 1, 8, 15, 22 Cycles 3-6: days 1, 15 Cycles 7+: day 1
  Lenalidomide: 25 mg/d on day 1-21 of every 28-day cycle.
  Dexamethasone: 40 mg/d on days 1, 8, 15, 22 of every 28-day cycle in participants < 75 years; 20 mg/d on days 1, 8, 15, 22 of every 28-day cycle in participants ≥ 75 years
  Interventions: Drug: Belantamab Mafodotin-Blmf; Drug: Daratumumab; Drug: Lenalidomide; Drug: Dexamethasone

INTERVENTIONS:
Drug: Belantamab Mafodotin-Blmf — Blmf will be available as 100 mg/vial in single-use vial for reconstitution, supplied as lyophilized powder.
  Blmf will be delivered as IV solution over at least 30 minutes.
Drug: Daratumumab — Daratumumab will be administered with subcutaneous injections. On days where Blmf is given together with daratumumab, daratumumab should be performed first.
Drug: Lenalidomide — Lenalidomide will be administered per os.
Drug: Dexamethasone — Dexamethasone will be administered intravenously or per os.

SUMMARY:
This is a phase 1/2, open label, study designed to assess the safety and clinical activity of different belantamab mafodotin doses in combination with daratumumab, lenalidomide and dexamethasone.

The study will evaluate different doses of belantamab mafodotin in combination with daratumumab, lenalidomide and dexamethasone in 2 cohorts and will determine the recommended phase 2 dose (RP2D) to be further evaluated for safety and clinical activity in the dose expansion cohort. The RP2D dose will be used for future studies in the transplant ineligible newly diagnosed multiple myeloma setting.

Overall, approximately 36 participants will be enrolled in the study. Participant follow-up will continue up to 3 years after the last participant is randomized. The estimated accrual period will be 12 months corresponding to an approximate total study duration of 4 years.

ELIGIBILITY:
Inclusion Criteria:

1. Participant must be ≥ 18 years or older.
2. Monoclonal plasma cells in the bone marrow ≥10% or presence of a biopsy proven plasmacytoma and documented MM satisfying at least one of the calcium, renal, anemia, bone (CRAB) criteria or biomarkers of malignancy criteria:

   CRAB criteria:

   v. Hypercalcemia: serum calcium >0.25 mmol/L (>1 mg/dL) higher than upper limit of normal (ULN) or >2.75 mmol/L (>11 mg/dL).

   vi. Renal insufficiency: creatinine clearance <40mL/min or serum creatinine >177 μmol/L (>2 mg/dL).

   vii. Anemia: hemoglobin >2 g/dL below the lower limit of normal or hemoglobin <10 g/dL.

   viii. Bone lesions: one or more osteolytic lesions on skeletal radiography, CT, or PET-CT.

   Biomarkers of Malignancy:

   d. Clonal bone marrow plasma cell percentage ≥60%. e. Involved: uninvolved serum free light chain (FLC) ratio ≥100. f. More than 1 focal lesion on magnetic resonance imaging (MRI) studies.
3. Must have at least ONE aspect of measurable disease, defined as one of the following:

   1. Urine M-protein excretion ≥200 mg/24 hrs (≥0.2 g/24 hrs), or
   2. Serum M-protein concentration ≥0.5 g/dL (≥5.0 g/L), or
   3. Serum FLC assay: involved FLC level ≥10 mg/dL (≥100 mg/L) and an abnormal serum FLC ratio (<0.26 or >1.65).
4. Not a candidate for high-dose chemotherapy with ASCT due to presence of significant comorbid condition(s), such as cardiac, pulmonary or other major organ dysfunction that are likely to have a negative impact on tolerability of high dose chemotherapy with stem cell transplantation. The participants will be assessed by the IMWG frailty index, a scoring system based on age, comorbidities and cognitive and physical conditions, which is recommended by the ESMO guidelines. Participants with IMWG frailty index score 1 or 2 will be considered transplant ineligible. The reason(s) for transplant ineligibility will be collected in the case report forms (CRFs).
5. ECOG performance status of 0-2 (see Appendix 1).
6. Adequate organ system function as defined by the below laboratory assessments. Hematologic

   1. Absolute neutrophil count (ANC) ≥1.25 X 109/L; GCSF use within the past 14 days are NOT permitted.
   2. Hemoglobin ≥ 8.0 g/dL; transfusions within the past 14 days are NOT permitted.
   3. Platelet count ≥ 50 x 109/L if bone marrow is >50% involved in myeloma. Otherwise ≥75 x 109/L; transfusions within the past 14 days are NOT allowed to reach this level.

      Hepatic
   4. Total bilirubin ≤1.5xULN (isolated bilirubin ≥1.5xULN is acceptable if bilirubin is fractionated and direct bilirubin <35%).
   5. ALT ≤ 2.5xULN. Renal
   6. eGFR ≥30 mL/min/1.73 m2; calculated using the Modified Diet in Renal Disease (MDRD) formula.
   7. Spot urine (albumin/creatinine ratio) <500 mg/g (56 mg/mmol) OR
   8. Urine Dipstick: Negative trace; if ≥1+ only eligible if confirmed <500 mg/g [56 mg/mmol] by albumin/creatinine ratio (spot urine from first void).
7. Female participants: contraceptive use should be consistent with local regulations regarding the methods of contraception for those participating in clinical studies:

   A female participant is eligible to participate if she is not pregnant or breastfeeding, and at least one of the following conditions applies:
   * Is not a woman of childbearing potential (WOCBP) defined as follows:

     1. ≥ 45 years of age and has not had menses for > 1 year
     2. Participants who have been amenorrhoeic for < 2 years without history of a hysterectomy and oophorectomy must have a follicle stimulating hormone value in the postmenopausal range upon screening evaluation
     3. Post-hysterectomy, post-bilateral oophorectomy, or post-tubal ligation. Documented hysterectomy or oophorectomy must be confirmed with medical records of the actual procedure or confirmed by an ultrasound. Tubal ligation must be confirmed with medical records of the actual procedure.

        OR
   * Is a WOCBP and using two methods of reliable birth control (one method that is highly effective and one additional effective [barrier] method), beginning 4 weeks before initiating treatment with lenalidomide, during therapy, during dose interruptions, and continuing for 4 weeks following discontinuation of lenalidomide treatment. Thereafter, WOCBP participants must use one method of reliable birth control that is highly effective for a further 4 months following discontinuation of belantamab mafodotin or 3 months following the discontinuation of daratumumab. WOCBP must also agree not to donate eggs (ova, oocytes) for the purpose of reproduction during treatment, during dose interruptions and for 28-days following the last dose of lenalidomide or 3 months following discontinuation of daratumumab treatment or 4 months following discontinuation of belantamab mafodotin treatment whichever is longer. For contraception guidance please refer to Appendix 2.

   A WOCBP must have two negative pregnancy tests before therapy initiation. The first test should be performed within 10-14 days and the second test within 24 hours before the start of lenalidomide therapy.

   The participant should not receive lenalidomide until the investigator has verified that the results of these pregnancy tests are negative. The investigator should evaluate the effectiveness of the contraceptive method in relationship to the first dose of study treatment. The investigator is responsible for a review of medical history, menstrual history, and recent sexual activity to decrease the risk for inclusion of a woman with a nearly undetected pregnancy.
8. Male participants: contraceptive use should be consistent with local regulations regarding the methods of contraception for those participating in clinical studies:

   Male participants are eligible to participate if they agree to the following during the intervention period and until 28 days after the last dose of lenalidomide or 3 months following the discontinuation of daratumumab or 6 months after the last dose of belantamab mafodotin, whichever is longer, to allow for clearance of any altered sperm.

   • Refrain from donating sperm

   PLUS either:
   * Be abstinent from heterosexual intercourse as their preferred and usual lifestyle (abstinent on a long term and persistent basis) and agree to remain abstinent, OR
   * Must agree to use contraception/barrier as detailed below:

   Agree to use a male condom, even if they have undergone a successful vasectomy, and female partner to use an additional highly effective contraceptive method with a failure rate of <1% per year as when having sexual intercourse with a woman of childbearing potential (including pregnant females).
9. Participants must be able to understand the study procedures and agree to participate in the study by providing written informed consent.

Exclusion Criteria:

Participants are excluded from the study if any of the following criteria apply:

1. Prior systemic therapy for MM, or SMM.

   * NOTE 1: An emergency course of steroids (defined as no greater than 40 mg of dexamethasone [or equivalent] per day for a maximum of 4 days [that is, a total of 160 mg]) is permitted.
   * NOTE 2: Focal palliative radiation is permitted prior to enrollment, provided that it occurred at least 2 weeks before the first dose of study drug, that the participant has recovered from radiation-related toxicities, and that the participant did not require corticosteroid administration (for a longer period than that specified in NOTE 1 above) for radiation-induced adverse events
2. Peripheral neuropathy or neuropathic pain Grade 2 or higher, as defined by the National Cancer Institute, Common Toxicity Criteria for Adverse Events (NCI CTCAE) Version 5.
3. Major surgery within 2 weeks before the first dose of study drug (NOTE: participant must be clinically stable following a major surgery to be entered in the study).
4. Presence of active renal condition (infection, requirement for dialysis, or any other significant condition that could affect participant's safety). Participants with isolated proteinuria resulting from MM are eligible, provided that they fulfil the other inclusion criteria.
5. Any serious and/or unstable pre-existing medical or psychiatric disorder, or other conditions (including laboratory abnormalities) that could interfere with participant's safety, obtaining informed consent, or compliance to the study procedures.
6. Evidence of active mucosal or internal bleeding uncontrolled by local therapy and not explained by reversible coagulopathy.
7. Current active unstable liver or biliary disease defined by the presence of ascites, encephalopathy, coagulopathy, hypoalbuminemia, esophageal or gastric varices, persistent jaundice, or cirrhosis. (except for Gilbert's syndrome or asymptomatic gallstones; otherwise stable non-cirrhotic chronic liver disease; or hepatobiliary involvement of malignancy as per the Investigator's assessment).
8. Participants with previous or concurrent malignancies other than MM are excluded. Exceptions are surgically treated cervical carcinoma in situ, or any other malignancy that has been considered medically stable for at least 2 years. The participant must not be receiving active therapy, other than hormonal therapy for this disease.

   o NOTE: Participants with curatively treated non-melanoma skin cancer are allowed without a 2-year restriction.
9. Evidence of cardiovascular risk including any of the following:

   * Evidence of current clinically significant untreated arrhythmias, including clinically significant ECG abnormalities, second degree (Mobitz Type II), or third degree atrioventricular (AV) block.
   * Screening 12-lead ECG showing a baseline QT interval >470 msec
   * History of myocardial infarction, acute coronary syndromes (including unstable angina), coronary angioplasty, or stenting or bypass grafting within 3 months of Screening.
   * Class III or IV heart failure as defined by the New York Heart Association functional classification system (Appendix 3).
   * Uncontrolled hypertension.
10. Participant has known chronic obstructive pulmonary disease (COPD) (defined as a forced expiratory volume in 1 second [FEV1] <50% of predicted normal), persistent asthma, or a history of asthma within the last 2 years (controlled intermittent asthma or controlled mild persistent asthma is allowed). NOTE: Participants with known or suspected COPD must have an FEV1 test at screening.
11. Active infection requiring treatment.
12. Known HIV infection, unless the participant can meet all of the following criteria:

    * Established anti-retroviral therapy (ART) for at least 4 weeks and HIV viral load <400 copies/mL.
    * CD4+ T-cell (CD4+) count ≥350 cells/uL.
    * No history of AIDS-defining opportunistic infections within the last 12 months. o NOTE: consideration must be given to ART and prophylactic antimicrobials that may have a drug:drug interaction and/or overlapping toxicities with belantamab mafodotin or other combination products as relevant (See Section 7.2, Drug Interactions)
13. To be seropositive for hepatitis B (defined by a positive test for hepatitis B surface antigen [HBsAg]) at screening or within 3 months prior to first dose of study treatment.

    * NOTE 1: Participants with resolved infection (i.e., participants who are positive for antibodies to hepatitis B core antigen [antiHBc] or antibodies to hepatitis B surface antigen [antiHBs]) must be screened using real-time polymerase chain reaction (PCR). Those who are PCR positive will be excluded.
    * NOTE 2: presence of antiHBs indicating previous vaccination will not constitute an exclusion criterion.
14. Positive hepatitis C antibody test result or positive hepatitis C RNA test result at screening or within 3 months before the first dose of study treatment unless the participant can meet the following criteria:

    * RNA test negative
    * Successful anti-viral treatment (usually 8 weeks duration) is required, followed by a negative hepatitis c virus (HCV) RNA test after a washout period of at least 4 weeks.
15. Current corneal epithelial disease except for mild punctate keratopathy.

    o NOTE: Participants with mild punctate keratopathy are allowed.
16. Intolerance or contraindications to anti-viral prophylaxis.
17. Unable to tolerate antithrombotic prophylaxis.
18. Active or history of venous thromboembolism within past 3 months.
19. AL amyloidosis (light chain amyloidosis), active POEMS syndrome (polyneuropathy, organomegaly, endocrinopathy, monoclonal plasma proliferative disorder, skin changes) or active plasma cell leukemia at the time of screening.
20. Exhibiting clinical signs of or with a known history of meningeal or central nervous system involvement by MM.
21. Known intolerance or immediate or delayed hypersensitivity reaction or idiosyncratic reaction to: drugs chemically related to belantamab mafodotin, or any of the components of the study treatment; daratumumab subcutaneous (SC) or to any of its excipients; or infused protein products, sucrose, histidine, and polysorbate 80.
22. Use of an investigational drug within 14 days or 5 half-lives (whichever is longer) preceding the first dose of study drug.
23. Plasmapheresis within 7 days before the first dose of study drug.
24. Participants with uncontrolled skin disease.
25. Participants with concomitant administration of a strong or moderate CYP3A4 inhibitor or inducer
26. Any serious and/or unstable pre-existing medical, psychiatric disorder or other conditions (including lab abnormalities) that could interfere with participant's safety, obtaining informed consent or compliance to the study procedures.
27. Participant must not have received a live or live-attenuated vaccine within 30 days prior to first dose of belantamab mafodotin.
28. Participant should not use contact lenses while receiving belantamab mafodotin.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2022-04-13 (Actual); Primary Completion 2026-03-15 (Estimated); Study Completion 2026-03-15 (Estimated)

PRIMARY OUTCOMES:
Part 1: Dose-Limiting Toxicity (DLT) | Up to 28 days
  The number (%) of participants and 95% CI with the DLT in each of the cohorts 1-2, using the DLT evaluable population.
Part 1 and 2: Adverse Events (AEs) and Serious adverse events (SAEs) | Up to 4 years
  The number (%) of participants with AEs and SAEs in each of the cohorts 1-2, using the DLT evaluable and Safety populations.
Part 1 and 2: Ocular toxicity | Up to 4 years
  Number of participants with ocular toxicity of Grade 2 or higher (per KVA scale).
Part 2: Overall Response Rate (ORR) | Up to 4 years
  ORR as per IMWG by Investigator assessment; defined as the percentage of participants with a confirmed partial response (PR), very good partial response (VGPR), complete response (CR) or stringent CR (sCR) (For the 'intention to treat' (ITT) population).

SECONDARY OUTCOMES:
Part 1: Overall Response Rate | Up to 4 years
  ORR and 95% CI as per IMWG by Investigator Assessment. ORR is defined as the percentage of participants with a confirmed PR, VGPR, CR or sCR.
Part 1 and 2: Lenalidomide Relative Dose Intensity (RDI) | Up to 4 years
  The RDI is defined as the percentage of the total administered over the total planned lenalidomide dose.
Part 1 and 2: Cumulative dose of belantamab mafodotin | Up to 4 years
  Cumulative belantamab mafodotin dose of (DLT evaluable population, safety population) administered in combination with daratumumab, lenalidomide and dexamethasone, i.e., the total dose of belantamab mafodotin that was administered.
Part 1: Very good partial response | Up to 4 years
  VGPR+ and 95% CI as per IMWG by Investigator Assessment (ITT population) [Part 1 only]; ORR is defined as the percentage of participants with a confirmed VGPR, CR or sCR.
Part 1 and 2: Time to response (TTR) | Up to 4 years
  TTR as per IMWG by Investigator Assessment (ITT population). TTR is defined as the time (in months) between the date of randomization and the first evidence of confirmed response (PR or better) for participants who achieve a response (i.e., confirmed PR or better).
  Descriptive methods will be used for the estimation of the time to response (i.e., mean, standard deviation, median, 1st and 3rd quartiles, minimum value and maximum value).
Part 1 and 2: Duration of response | Up to 4 years
  DoR as per IMWG by Investigator Assessment (ITT population). DoR is defined as the time (months) from first evidence of confirmed PR or better until the earliest date of: documented disease progression (PD) per IMWG response criteria; or death due to PD among participants who achieved a response of PR or better. For alive and progression-free participants, data will be censored at the date of initiation of the subsequent line of treatment or at the last date of follow-up that the participant was known to be alive and progression-free.
  The Kaplan-Meier method will be used for the estimation of DoR. The median DoR will be presented along with the respective 95% confidence intervals [CIs]) and the 1st and 3rd quartiles.
Part 1 and 2: Complete response rate (CRR) | Up to 4 years
  CRR as per IMWG by Investigator Assessment (ITT population). CRR is defined as the percentage of participants with a confirmed CR or sCR. The denominator will be the total number of participants in each population, cohort and group respectively.
Part 1 and 2: Minimal residual disease (MRD) negativity rate | Up to 4 years
  MRD negativity rate (ITT population) is defined as the number (%) of participants who achieve MRD negativity (at or below the threshold of 10-5), assessed via Next Generation Flow (NGF). The denominator will be the total number of participants in each population, cohort and Group respectively.
Part 1 and 2: Progression free survival (PFS) | Up to 4 years
  PFS as per IMWG by Investigator Assessment (ITT population, Safety population). PFS is defined as the time (in months) from randomization until the earliest date of documented PD per IMWG, or death due to any cause. For participants who neither progress nor die, the PFS will be censored at the date of their last adequate disease assessment. For participants who start a new anti-myeloma treatment, PFS will be censored at the date of the last adequate assessment before the start of the new treatment. For a randomized participant who does not have any post-baseline disease assessments and who has not died, PFS will be censored at the randomization date.
  The median PFS will be analyzed with the Kaplan Meier method and presented along with the respective 95% CI and the 1st and 3rd quartiles.
Part 1 and 2: Overall survival (OS) | Up to 4 years
  OS is defined as the time from first dose/randomization until death due to any cause. If a participant is not known to have died, survival time will be censored at the date of last contact ("last known date alive").
  The median OS will be analyzed using the Kaplan-Meier method and will be presented with the respective 95% CI and the 1st and 3rd quartiles.
Part 1 and 2: Abnormal ocular findings | Up to 4 years
  Number (%) of participants with abnormal ocular findings (on ophthalmic exam) (DLT evaluable population, Safety population).
Part 1 and 2: Pharmacokinetics (PK) analysis (PK population) - Peak plasma Concentration (Cmax) | Up to 4 years
  Concentration-time data: linear and semi-logistic unique profiles of concentration-time and the mean and median profiles (as applicable) will be graphically represented for belantamab mafodotin. Belantamab mafodotin concentrations will be presented for each participant and summarized (as applicable) at each PK timepoint and cohort.
  PK parameters: Concentration-time data can be presented, considering data from other studies and analyzed using a population PK analysis. The Cmax will be calculated. The results of these analyses can be included in a separate report.
  PK parameters will be descriptively summarized using mean, median, standard deviation (SD), and 95% CI, minimum/maximum value, geometric mean and coefficient of variation.
Part 1 and 2: PK analysis (PK population) - Area under the plasma concentration versus time curve (AUC) | Up to 4 years
  Concentration-time data: linear and semi-logistic unique profiles of concentration-time and the mean and median profiles (as applicable) will be graphically represented for belantamab mafodotin. Belantamab mafodotin concentrations will be presented for each participant and summarized (as applicable) at each PK timepoint and cohort.
  PK parameters: Concentration-time data can be presented, considering data from other studies and analyzed using a population PK analysis. The AUC will be calculated. The results of these analyses can be included in a separate report.
  PK parameters will be descriptively summarized using mean, median, standard deviation (SD), and 95% CI, minimum/maximum value, geometric mean and coefficient of variation.
Part 1 and 2: Ocular Surface Disease Index (OSDI) | Up to 4 years
  Number of participants with changes from baseline and proportion of participants with within-participant meaningful change in self reported ocular symptoms and related impacts as measured by the OSDI questionnaire.
Part 1 and 2: Alternate corneal AE management | Up to 4 years
  KVA events, dose holds, worst post-baseline BCVA and incidence of Grade 4 corneal findings will be descriptively summarized using frequencies and proportions. No statistical comparison will be made between the 2 groups.

CONTACTS AND LOCATIONS:
Overall Officials: Evangelos Terpos, Prof, Principal Investigator — Department of Clinical Therapeutics, School of Medicine, National Kapodistrian University of Athens (NKUA)
Locations (2):
- Greece (2):
  - Department of Clinical Therapeutics, School of Medicine, National Kapodistrian University of Athens (NKUA), Athens
  - Anticancer Hospital of Thessaloniki "Theageneio", Thessaloniki

IPD SHARING:
Plan to Share IPD: No